CLINICAL TRIAL: NCT01702753
Title: Bifidobacterium Animalis Subsp. Lactis in Prevention of Common Infections in Healthy Children Attending Day Care Centers - Randomized, Double Blind, Placebo Controlled Study
Brief Title: Bifidobacterium Animalis Subsp. Lactis in Prevention of Common Infections in Healthy Children Attending Day Care Centers
Acronym: PROBBIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Zagreb (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROBBIC I Study
Record Dates: First submitted 2012-10-03; First posted 2012-10-08 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Gastrointestinal Tract Infections; Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bifidobacterium animalis subsp. lactis (Active Comparator)
  Interventions: Dietary Supplement: Bifidobacterium animalis subsp. lactis
- Placebo (Placebo Comparator)

INTERVENTIONS:
Dietary Supplement: Bifidobacterium animalis subsp. lactis
  Arms: Bifidobacterium animalis subsp. lactis

SUMMARY:
Hypothesis: Use of Bifidobacterium animalis subsp. lactis can effectively prevent common infections (gastrointestinal and respiratory) in healthy children who attend day care centre

This study is a prospective, randomized, double blind, placebo- controlled parallel study in healthy children attending day care centers.

The study will investigate the effect of supplementation with the probiotic strain Bifidobacterium animalis subsp. lactis on the incidence and duration of gastrointestinal and respiratory infections and absence from day care due to infections.

The test product is a sachet containing 1 gram of powder. The test product will contain minimum 1 billion CFU (colony forming units) of probiotic per serving. The placebo product is an identical product except for the absence of probiotics.

The study includes 3 months (90 days) of intervention period. The study product will be consumed daily in the evening together with a meal.

The consumption of the study products will be taken under the surveillance of the parents.

During the entire intervention period the subjects are not allowed to consume any probiotic products other than the study products supplied to them by the study personnel.

Data on infections will be recorded in a diary, filled in and administered by the parents and diary recorded by referring physician (on-call log).

All infections are to be diagnosed by the local physician. The incidence of infections will be analyzed based on the information recorded in the diaries (parent's & physician's).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children attending day care at kindergartens located in the Zagreb's city centre
* Age from 1 year to 7 years
* Attendance at daycare centers: > 3 days per week
* Signed informed consent by the parents

Exclusion Criteria:

* Immunodeficiency
* Receiving probiotic and /or prebiotic products prior to enrolment (2 weeks prior to study start)
* Neoplasms
* Severe chronic disorders

Ages: 1 Year to 7 Years | Sex: All
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Common infections
  Number of children with gastrointestinal tract infections defined as diarrhoea (3 or more loose or watery stools in 24 hours or increase of number of stools for more than 50% in 24 hours) or vomiting (defined by physician and not a result of other symptoms including cough or diseases including gastroesophageal reflux disease or neurological conditions) or both.
  And number of children with respiratory tract infections defined as: pharyngitis, otitis, common cold, pneumonia, bronchitis and bronciolitis (all infections diagnosed by physician) Number of children with adverse events.

SECONDARY OUTCOMES:
Duration of symptoms
  Duration of symptoms in days

OTHER OUTCOMES:
Infections with determined infective cause
  Number of gastrointestinal and erspiratory tract infections with proven infective cause (if determined)

CONTACTS AND LOCATIONS:
Locations (1):
- Djecji vrtic Matija Gubec, Zagreb, Croatia

REFERENCES:
- [Derived] Hojsak I, Mocic Pavic A, Kos T, Dumancic J, Kolacek S. Bifidobacterium animalis subsp. lactis in prevention of common infections in healthy children attending day care centers - Randomized, double blind, placebo-controlled study. Clin Nutr. 2016 Jun;35(3):587-91. doi: 10.1016/j.clnu.2015.05.004. Epub 2015 May 19. PMID 26031908